CLINICAL TRIAL: NCT06487169
Title: Effectivity of the Air Extraction to Prevent Anesthesiologists Waste Anesthetic Gas Exposure of Sevoflurane During Pediatric Induction
Brief Title: Effectivity Gas Extraction to Prevent Anesthesiologists Waste Gas Exposure of Sevofluorane During Pediatric Induction
Status: Not yet recruiting | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MOSTAFA.SOMRI, Clinical Associate Professor, Bnai Zion Medical Center
Other Study IDs: 0072-24-BNZ
Record Dates: First submitted 2024-06-24; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Unrecognized Condition
Keywords: sevofluorane,; hexacloroisopropanolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Anesthesiologists
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urine analysis to determine the presence of hexafluoroisopropanol — analysis of sevoflurane metabolites in urine

SUMMARY:
Inhalational anesthetics (IAs) are widely used in surgery and experimental research. IAs, in addition to their medical significance, are a major source of chemical contamination in the operating rooms (ORs).Exposure to IAs in ORs personnel results in reproductive effects, including infertility , spontaneous abortions , congenital diseases , psychological and neurological disturbances, hepatotoxicity , and genotoxicity .The metabolites of sevoflurane include hexafluoroisopropanol (HFIP) and inorganic fluoride (IF). The hospital's engineering department installed an air extractor with the objective to reduce the anesthetic gas concentrations during pediatric anesthesia induction. The investigators are interested in checking if the new technique also has an influence in decreasing the level of Sevoflurane breathed in by the anesthesiologist.The investigators purpose is to detect the presence of desfluoroisopropanolol in the urine of ten anesthesiologists who used sevoflurane to induce children with a mask during an eight-hour session in the induction room (IR) One session will be conducted without the use of the air extractor and the other with the air extractor. After 24 hours, a urine sample will be taken and sent to the Toxicology Unit.

DETAILED DESCRIPTION:
IAs are widely used in surgery. IAs, in addition to their medical significance, are a major source of chemical contamination in the ORs, dental clinics, delivery rooms, and intensive care units Although ORs are equipped with ventilation and scavenging systems, it should be noted that occupational exposure to IAs is still higher than threshold limit value recommended by Occupational Safety and Health Administration (OSHA) .

Exposure to IAs in ORs personnel results in 1. reproductive effects, including 2. infertility 3., spontaneous abortions 4., congenital diseases 5., psychological and neurological disturbances 6., hepatotoxicity 7., and genotoxicity 8.

Possible mechanisms underlying the genotoxic effects of these agents are not clear. It seems that oxidative stress through excessive production of reactive oxygen species (ROS), including superoxide, hydroxyl, and hydrogen peroxide is an important mechanism by which ionizing radiation and IAs cause DNA damage 8.

Urinary HFIP has been recently suggested as a valuable biomarker for the monitoring of occupational exposure of medical staff exposed to low concentration of airborne sevoflurane in operating rooms Minimizing the impact of anesthetic gases contributes to the protection of individuals who experience chronic risk of occupational exposure from waste gases in working environments with poor or inadequate scavenging of inhaled anesthetics.

To ensure occupational safety around IAs in 1977, the US National Institute for Occupational Safety and Health (NIOSH) recommended that occupational exposure to halogenated anesthetics agents should not exceed 2 ppm or N2O >25 ppm within a 1-hour period (reweighted average for exposure duration) To manage and minimize occupational exposure to WAGs, NIOSH and others highlight the pivotal importance of using an efficient air ventilation Anesthesia induction specially a performed with needle injection is a stressful part of surgery for pediatric patients and their parents. Children may undergo physical, mental, and physiological distress due to anxiety at the time of induction and after surgery, and higher parental anxiety levels are directly associated with children's preoperative anxiety levels .

The parental presence during the use of facial mask to performed the induction with IAs contribute significantly to reduce the anxiety in the children's.

In the Anesthesiology Department of the Bnai Zion Medical Center, the induction technique is performed with sevofluorane and Nitrous Oxide gas loaded through a mask and with parenteral presence.

This anesthetic approach demands to use the mask to perform the induction, therefore, it is not adapted closely to the face of the patient during the short period of time when the child is in the excitatory face. During this time, part of the fresh gas supply leaks to the air of the Pediatric Induction Room (PIR). This technique obviously increases the concentration of sevoflurane and Nitrous Oxide( N2O) over the safety recommended standards range.

In 2022 measurements in a PIR revealed sevoflurane concentrations far above safety standards of 1 to 2 ppm reaching as high as 33.4 ppm. and measurements of N2O concentrations exceeding safety standards of 25 ppm, reaching values as high as 125 ppm .

Since the PIR is not equipped with an air extraction system, the hospital's engineering department installed an air extractor with the objective to reduce the anesthetic gas concentrations during pediatric anesthesia induction.

The investigators checked the levels of sevoflurane in the air of the induction room without the removal of air with sevoflurane and with the removal of air contaminated with sevoflurane.

The average sevoflurane concentration recorded without use of the air extractor was (Mean = 10.86, SD = 8.67) significantly exceeded the mean concentration of sevoflurane observed subsequent to the extractor application (Mean = 0.18, SD = 0.31) Stimulated by the results obtained in the PIR air, we are interested in checking if the new technique also has an influence in decreasing the level of Sevoflurane breathed in by the anesthesiologist.

HFIP is a major metabolite of sevoflurane and is excreted in the urine within the first few hours after exposure.

The Laboratory of Clinical Toxicology, Pharmacology and Pharmacogenetic of the Rambam Health Care Campus has the capability to identifying and quantifying the HFIP in urine using the technique of Mass Spectrometry.

The investigators purpose is to detect the presence of HFIP in the urine of ten anesthesiologists who used sevoflurane to induce children with a mask during an eight-hour session in the PIR. One session will be conducted without the use of the air extractor and the other with the air extractor. After 24 hours, a urine sample will be taken and sent to the Toxicology Unit.

ELIGIBILITY:
Inclusion Criteria: anesthesiologists that work in pediatric anesthesia room performed induction anesthesia with sevoflurane delivery by mask -

Exclusion Criteria: anesthesia that required IV induction and that not use sevoflurane

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ten anesthesiologists that work in Pediatric Induction Room using anesthesia induction with sevoflurane delivery with mask
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Presence of sevoflurane metabolite, hexafluoroisopropanol in urine | up to 24 weeks
  hexafluoroisopropanol is the metabolism of the sevofluorane